CLINICAL TRIAL: NCT02735044
Title: 6-Month, Multicenter, Randomized, Open-label, 2-Arm, Parallel-group Study Comparing the Efficacy and Safety of a New Formulation of Insulin Glargine and Lantus® Injected Once Daily in Children and Adolescents Age 6 - 17 Years With Type 1 Diabetes Mellitus With a 6-month Safety Extension Period
Brief Title: Comparison of the Safety and Efficacy of HOE901-U300 With Lantus in Children and Adolescents With Type 1 Diabetes Mellitus
Acronym: EDITION JUNIOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC13957; 2015-002084-42 (EudraCT Number); U1111-1168-4546 (Other: UTN)
Record Dates: First submitted 2016-03-30; First posted 2016-04-12 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOE901-U300 (Experimental): HOE901-U300 (Insulin glargine 300 Units/milliliter [U/mL]) Subcutaneous(SC) injection once daily for 12 months.
  Interventions: Drug: Insulin glargine,300 U/mL; Drug: Background therapy
- Lantus (Active Comparator): Lantus (Insulin glargine 100 U/mL) SC injection once daily for 12 months.
  Interventions: Drug: Insulin glargine (100 units /mL); Drug: Background therapy

INTERVENTIONS:
Drug: Insulin glargine,300 U/mL — Subcutaneous injection in the morning or evening using a prefilled pen. Dose titration to achieve fasting self-monitored plasma glucose (SMPG) from 90 to 130 milligram/deciliter (mg/dL) (5.0 to 7.2 millimol per liter [mmol/L])
  Other Names: Toujeo ®
  Arms: HOE901-U300
Drug: Insulin glargine (100 units /mL) — Subcutaneous injection in the morning or evening using a prefilled pen. Dose titration to achieve fasting SMPG from 90 to 130 mg/dL (5.0 to 7.2 mmol/L)
  Arms: Lantus
Drug: Background therapy — Fast-acting mealtime insulin analogs

SUMMARY:
Primary Objective:

To compare the efficacy of a new formulation of insulin glargine (HOE901-U300) to Lantus in terms of change of HbA1c from baseline to endpoint (month 6) in children and adolescents with type 1 diabetes mellitus.

.

Secondary Objectives:

To compare HOE901-U300 and Lantus in terms of:

* Percentage of participants reaching target HbA1c and fasting plasma glucose (FPG).
* To assess the safety of HOE901-U300 including analysis of events of hypoglycemia, events of hyperglycemia with ketosis, and development of anti-insulin-antibodies.

DETAILED DESCRIPTION:
The study duration per participant was approximately 58 weeks that consisted of a 2 week screening period, a main 6-month comparative efficacy and safety treatment period, a 6-month comparative safety extension period, and a 4-week post treatment follow up period.

ELIGIBILITY:
Inclusion criteria :

* Children and adolescents with type 1 diabetes mellitus (T1DM) for at least 1 year confirmed by typical symptoms at diagnosis and/or by antibody testing [presence of anti-GAD (glutamic acid decarboxylase) or anti-IA2 (islet antigen 2/tyrosine phosphatase) or anti-islet cell antibodies] and/or clinical features (eg, history of ketoacidosis)].
* Signed written informed consent obtained from parent(s)/legal guardian and written or oral assent obtained from participant.

Exclusion criteria:

* Age <6 years and >=18 years at randomization.
* Less than 1 year on insulin treatment prior to screening visit.
* Less than 6 months on basal plus mealtime insulin and self-monitoring of blood glucose prior to screening visit.
* Participants using premix insulins in the last 3 months before screening visit or participants using human regular insulin as mealtime insulin in the last 3 months before screening visit.
* Use of an insulin pump in the last 6 months before screening visit or plans to switch to pump within the next 6 months after screening visit.
* Any contraindication to use of insulin glargine as defined in the national product label.
* No willingness to inject insulin glargine (Lantus or HOE901-U300) once daily.
* HbA1c <7.5% or >11% at screening.
* Initiation of any glucose-lowering medications in the last 3 months before screening visit.
* Hospitalization or care in the emergency ward for diabetic ketoacidosis or history of severe hypoglycemia (as defined by need for glucagon or IV glucose) and accompanied by seizure and/or unconsciousness and/or coma in the last 3 months prior to screening visit.
* Postmenarchal girls not protected by highly-effective method(s) of birth control and/or who were unwilling or unable to be tested for pregnancy. Abstinence from sexual intercourse was considered as an acceptable form of birth control.
* Pregnant or breast-feeding adolescents, or adolescents who intended to become pregnant during the study period, or who were at risk of getting pregnant due to any psychosocial reason during the study period.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 463 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (107):
- United States (13):
  - Investigational Site Number 8400008, Tucson, Arizona
  - Investigational Site Number 8400037, Atlanta, Georgia
  - Investigational Site Number 8400032, Indianapolis, Indiana
  - Investigational Site Number 8400015, Buffalo, New York
  - Investigational Site Number 8400016, Chapel Hill, North Carolina
  - Investigational Site Number 8400035, Morehead City, North Carolina
  - Investigational Site Number 8400038, Oklahoma City, Oklahoma
  - Investigational Site Number 8400030, Philadelphia, Pennsylvania
  - Investigational Site Number 8400010, Rapid City, South Dakota
  - Investigational Site Number 8400005, Dallas, Texas
  - Investigational Site Number 8400021, Dallas, Texas
  - Investigational Site Number 8400029, Lufkin, Texas
  - Investigational Site Number 8400034, Seattle, Washington
- Argentina (7):
  - Investigational Site Number 0320003, Caba
  - Investigational Site Number 0320001, Caba
  - Investigational Site Number 0320004, Capital Federal
  - Investigational Site Number 0320002, Capital Federal
  - Investigational Site Number 0320006, Mendoza
  - Investigational Site Number 0320005, Salta
  - Investigational Site Number 0320007, San Miguel de Tucumán
- Brazil (6):
  - Investigational Site Number 0760005, Curitiba
  - Investigational Site Number 0760006, Fortaleza
  - Investigational Site Number 0760004, Fortaleza
  - Investigational Site Number 0760003, Porto Alegre
  - Investigational Site Number 0760001, São Paulo
  - Investigational Site Number 0760002, São Paulo
- Bulgaria (3):
  - Investigational Site Number 1000001, Plovdiv
  - Investigational Site Number 1000005, Sofia
  - Investigational Site Number 1000004, Varna
- Canada (4):
  - Investigational Site Number 1240003, Halifax
  - Investigational Site Number 1240002, Montreal
  - Investigational Site Number 1240005, Montreal
  - Investigational Site Number 1240006, Sherbrooke
- Chile (5):
  - Investigational Site Number 1520002, Santiago
  - Investigational Site Number 1520004, Santiago
  - Investigational Site Number 1520006, Santiago
  - Investigational Site Number 1520007, Temuco
  - Investigational Site Number 1520003, Viña del Mar
- Czechia (3):
  - Investigational Site Number 2030003, Hradec Králové
  - Investigational Site Number 2030005, Ostrava - Poruba
  - Investigational Site Number 2030001, Praha 5 - Motol
- Investigational Site Number 2080001, Herlev, Denmark
- France (2):
  - Investigational Site Number 2500003, Montpellier
  - Investigational Site Number 2500002, Toulouse
- Germany (4):
  - Investigational Site Number 2760002, Hanover
  - Investigational Site Number 2760001, Heidelberg
  - Investigational Site Number 2760004, Leipzig
  - Investigational Site Number 2760003, Münster
- Hungary (7):
  - Investigational Site Number 3480001, Budapest
  - Investigational Site Number 3480004, Budapest
  - Investigational Site Number 3480003, Budapest
  - Investigational Site Number 3480005, Gyula
  - Investigational Site Number 3480002, Miskolc
  - Investigational Site Number 3480006, Pécs
  - Investigational Site Number 3480007, Székesfehérvár
- Israel (4):
  - Investigational Site Number 3760003, Beersheba
  - Investigational Site Number 3760001, Haifa
  - Investigational Site Number 3760006, Holon
  - Investigational Site Number 3760002, Petah Tikva
- Italy (5):
  - Investigational Site Number 3800001, Florence
  - Investigational Site Number 3800005, Roma
  - Investigational Site Number 3800004, Torino
  - Investigational Site Number 3800006, Varese
  - Investigational Site Number 3800003, Verona
- Japan (6):
  - Investigational Site Number 3920006, Chiyoda-Ku
  - Investigational Site Number 3920002, Fukuoka
  - Investigational Site Number 3920003, Hiroshima
  - Investigational Site Number 3920007, Kobe
  - Investigational Site Number 3920005, Osaka
  - Investigational Site Number 3920004, Shinjuku-Ku
- Latvia (2):
  - Investigational Site Number 4280002, Daugavpils
  - Investigational Site Number 4280001, Riga
- Mexico (5):
  - Investigational Site Number 4840003, Durango
  - Investigational Site Number 4840004, México
  - Investigational Site Number 4840001, Monterrey
  - Investigational Site Number 4840002, Puebla City
  - Investigational Site Number 4840005, Veracruz
- Investigational Site Number 8070001, Skopje, North Macedonia
- Poland (6):
  - Investigational Site Number 6160005, Bielsko-Biala
  - Investigational Site Number 6160001, Gdansk
  - Investigational Site Number 6160006, Szczecin
  - Investigational Site Number 6160007, Warsaw
  - Investigational Site Number 6160004, Warsaw
  - Investigational Site Number 6160003, Warsaw
- Romania (5):
  - Investigational Site Number 6420005, Bucharest
  - Investigational Site Number 6420007, Constanța
  - Investigational Site Number 6420004, Craiova
  - Investigational Site Number 6420006, Sibiu
  - Investigational Site Number 6420003, Timișoara
- Russia (4):
  - Investigational Site Number 6430001, Moscow
  - Investigational Site Number 6430002, Saint Petersburg
  - Investigational Site Number 6430004, Smolensk
  - Investigational Site Number 6430003, Ufa
- Serbia (3):
  - Investigational Site Number 6880002, Belgrade
  - Investigational Site Number 6880003, Belgrade
  - Investigational Site Number 6880004, Niš
- Spain (6):
  - Investigational Site Number 7240005, Barcelona
  - Investigational Site Number 7240002, Barcelona
  - Investigational Site Number 7240003, Esplugues de Llobregat
  - Investigational Site Number 7240004, Sabadell
  - Investigational Site Number 7240006, Santa Cruz de Tenerife
  - Investigational Site Number 7240001, Vitoria-Gasteiz
- Investigational Site Number 7520002, Stockholm, Sweden
- United Kingdom (4):
  - Investigational Site Number 8260005, Doncaster
  - Investigational Site Number 8260001, Ipswich
  - Investigational Site Number 8260004, Kettering
  - Investigational Site Number 8260002, Salisbury

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Danne T, Tamborlane WV, Malievsky OA, Franco DR, Kawamura T, Demissie M, Niemoeller E, Goyeau H, Wardecki M, Battelino T. Efficacy and Safety of Insulin Glargine 300 Units/mL (Gla-300) Versus Insulin Glargine 100 Units/mL (Gla-100) in Children and Adolescents (6-17 years) With Type 1 Diabetes: Results of the EDITION JUNIOR Randomized Controlled Trial. Diabetes Care. 2020 Jul;43(7):1512-1519. doi: 10.2337/dc19-1926. Epub 2020 May 19. PMID 32430458

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 105 centers in 24 countries. A total of 616 participants were screened between 14 April 2016 and 31 October 2017, of which 153 were screen failures. Screen failures were mainly due to glycated hemoglobin (HbA1c) level outside of defined ranges per eligibility criteria.
Pre-assignment Details: A total of 463 participants were randomized in the study. Randomization was stratified by age group (<12 years and >=12 years) and by HbA1c (<8.5% and >=8.5%). Assignment to arms was done centrally using interactive voice system in 1:1 ratio.
Groups:
- HOE901-U300: Insulin glargine 300 Units/milliliter (U/mL) subcutaneous (SC) injection once daily in the morning or evening for 12 months.
- Lantus: Insulin glargine 100 U/mL SC injection once daily in the morning or evening for 12 months.
Period: Overall Study
Arm/Group | HOE901-U300 | Lantus
Started | 233 | 230
Treated | 233 | 228
Completed | 217 | 207
Not Completed | 16 | 23
Not completed — Adverse Event | 3 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Poor compliance to protocol | 7 | 7
Not completed — Randomized and not treated | 0 | 2
Not completed — Other, not specified above | 5 | 11

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- HOE901-U300: Insulin glargine 300 U/mL SC injection once daily in the morning or evening for 12 months.
- Total: Total of all reporting groups
Arm/Group | HOE901-U300 | Lantus | Total
Number analyzed (Participants) | 233 | 230 | 463
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.9 (2.9) | 12.9 (2.9) | 12.9 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 121 | 226
  Male | 128 | 109 | 237
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Here, number analyzed = participants with available data for specified measure.
  Participants
    number analyzed (Participants) | 232 | 226 | 458
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 11 | 6 | 17
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 8 | 6 | 14
    White | 211 | 211 | 422
    More than one race | 2 | 2 | 4
    Unknown or Not Reported | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: BMI percentile] | 67.52 (26.62) | 69.13 (26.64) | 68.32 (26.61)
Hemoglobin A1C (HbA1C) [Mean (Standard Deviation); unit: percentage of A1C] | 8.65 (0.88) | 8.61 (0.87) | 8.63 (0.88)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c to Month 6
Description: Change in HbA1c was calculated by subtracting baseline value from Month 6 value. Adjusted least-square (LS) means and standard errors (SE) were obtained using analysis of covariance (ANCOVA) after multiple imputations of missing data using post-baseline HbA1c data available on the main 6-month randomized period.
Time Frame: Baseline to Month 6
Population: Analysis was performed on intent-to-treat (ITT) population that included all randomized participants, regardless of whether the treatment kit was used, and was analyzed according to the allocated treatment group. Here, 'Overall number of participants analyzed' signified number of participants with available data for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 232 | 230
Percentage of HbA1c | -0.399 (0.063) | -0.402 (0.064)
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; Analysis was performed using ANCOVA models which included the treatment group, the randomization stratum of age group at screening visit (<12 years and >=12 years), and the continuous fixed covariates of the baseline HbA1c value; Test type: Non-Inferiority — Non-inferiority of HOE901-U300 versus Lantus was demonstrated if the upper bound of the two-sided 95% confidence interval (CI) for the difference in the mean change in HbA1c from baseline to month 6 was <0.3%; LS Mean difference = 0.004, 95% CI 2-sided [-0.172 to 0.179], Standard Error of Mean 0.090
Statistical Analysis 2: Comparison: HOE901-U300 vs Lantus; A step-wise closed testing approach was used to control the type I error. Analysis was performed using ANCOVA models which included the treatment group, the randomization stratum of age group at screening visit (<12 years and >=12 years), and the continuous fixed covariates of the baseline HbA1c value; Test type: Superiority — Superiority of HOE901-U300 versus Lantus was demonstrated if the upper bound of the two-sided 95% CI for the difference between treatment groups was <0 (zero); p = 0.965, ANCOVA — Threshold for significance at 0.025 level

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) to Month 6
Description: Change in FPG was calculated by subtracting baseline value from Month 6 value. Adjusted LS means and SE were obtained using ANCOVA after multiple imputation to address missing data in the main 6 month randomized period.
Time Frame: Baseline to Month 6
Population: Analysis was performed on ITT population. Here, 'Overall number of participants analyzed' signified number of participants with available data for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 232 | 230
millimole per liter (mmol/L) | -0.563 (0.372) | -0.549 (0.372)

3. Secondary Outcome: Percentage of Participants With HbA1c Values of <7.5% at Month 6
Description: Participants without any available HbA1c assessment at month 6 and/or with a premature study discontinuation during the main 6-month randomized period were considered as a failure (non-responders) in the analysis. Analysis was performed using Cochran-Mantel-Haenszel (CMH) method with randomization strata of screening HbA1c (<8.5%; >=8.5%) and randomization strata of age at screening (<12 years, >=12 years).
Time Frame: Month 6
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 233 | 230
percentage of participants | 26.18 | 23.48

4. Secondary Outcome: Percentage of Participants With HbA1c Values of <7.5% Without Any Episode of Severe and/or Documented Self-Monitored Plasma Glucose ([SMPG] <54 mg/dL [3.0 mmol/L]) Symptomatic Hypoglycemia During the Last 3 Months of the Main 6-month Randomized Period
Description: as for outcome 3
Time Frame: upto Month 6
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 233 | 230
percentage of participants | 4.29 | 4.78

5. Secondary Outcome: Percentage of Participants With FPG of <=130 mg/dL (7.2 mmol/L) at Month 6
Description: Participants without any available FPG assessment at month 6 and/or with a premature study discontinuation during the main 6-month randomized period were considered as a failure (non-responders) in the analysis. Analysis was performed using Cochran-Mantel-Haenszel (CMH) method with randomization strata of screening HbA1c (<8.5%; >=8.5%) and randomization strata of age at screening (<12 years, >=12 years).
Time Frame: Month 6
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 233 | 230
percentage of participants | 27.47 | 26.52

6. Secondary Outcome: Percentage of Participants With FPG of <=130 mg/dL (7.2 mmol/L) Without Any Episode of Severe and/or Documented (SMPG <54 mg/dL [3.0 mmol/L]) Symptomatic Hypoglycemia During the Last 3 Months of the Main 6-month Randomized Period
Description: as for outcome 3
Time Frame: upto Month 6
Population: Analysis was performed on ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 233 | 230
percentage of participants | 9.44 | 7.39

7. Secondary Outcome: Change From Baseline in 24-Hour Mean Plasma Glucose Based on 8-point SMPG Profiles to Month 6
Description: 8-point SMPG profiles were measured at the following 8 points: between 01:00 and 04:00 (clock time) at night, pre-breakfast, 2 hours after breakfast, pre-lunch, 2 hours after lunch, pre-dinner, 2 hours after dinner, and bedtime. Analysis was performed using a ANCOVA model including the fixed categorical effects of treatment group, randomization strata of screening HbA1c (<8.5%; >=8.5%), randomization strata of age at screening (<12 years, >=12 years) and the baseline 24-hour average 8-point profile SMPG.
Time Frame: Baseline to Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 147 | 146
mmol/L | 0.139 (0.249) | -0.266 (0.250)

8. Secondary Outcome: Change From Baseline in Variability of 24-Hour Mean Plasma Glucose Based on 8-point SMPG Profiles at Month 6
Description: 8-point SMPG profiles were measured at the following 8 points: between 01:00 and 04:00 (clock time) at night, pre-breakfast, 2 hours after breakfast, pre-lunch, 2 hours after lunch, pre-dinner, 2 hours after dinner, and bedtime. Variability was assessed by the coefficient of variation (standard deviation divided by mean) calculated over the 8-point SMPG. Analysis was performed using a ANCOVA model including the fixed categorical effects of treatment group, randomization strata of screening HbA1c (<8.5%; >=8.5%) and randomization strata of age at screening (<12 years, >=12 years).
Time Frame: Baseline, Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of mean variability
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 147 | 146
percentage of mean variability | 1.469 (1.409) | 0.789 (1.415)

9. Secondary Outcome: Change From Baseline to Month 6 in 8-Point SMPG Profile Per Time Point
Description: 8-point SMPG profiles were measured for following 8 time points at Baseline and Month 6: between 01:00 and 04:00 (clock time) at night, pre-breakfast, 2 hours after breakfast, pre-lunch, 2 hours after lunch, pre-dinner, 2 hours after dinner, and bedtime.
Time Frame: Baseline to Month 6
Population: Analysis was performed on ITT population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 233 | 230
mmol/L
  Between 01:00 and 04:00 at night: number analyzed (Participants) | 109 | 116
  Between 01:00 and 04:00 at night | 0.84 (6.94) | -0.60 (7.08)
  Pre-breakfast: number analyzed (Participants) | 141 | 142
  Pre-breakfast | -0.41 (5.48) | -1.71 (6.56)
  2 hours after breakfast: number analyzed (Participants) | 135 | 128
  2 hours after breakfast | -0.26 (7.18) | -0.62 (6.78)
  Pre-lunch: number analyzed (Participants) | 144 | 140
  Pre-lunch | 0.43 (6.99) | 1.11 (6.85)
  2 hours after lunch: number analyzed (Participants) | 131 | 129
  2 hours after lunch | 0.49 (7.64) | -0.55 (7.20)
  Pre-dinner: number analyzed (Participants) | 141 | 136
  Pre-dinner | 0.29 (8.05) | -0.02 (6.78)
  2 hours after dinner: number analyzed (Participants) | 125 | 124
  2 hours after dinner | 0.51 (8.53) | 0.60 (6.86)
  Bedtime: number analyzed (Participants) | 114 | 117
  Bedtime | 0.86 (7.60) | -0.60 (7.00)

10. Secondary Outcome: Percentage of Participants With at Least One Hypoglycemic Events (Any Hypoglycemia, Severe Hypoglycemia, Documented Symptomatic, Probable Symptomatic, Asymptomatic Hypoglycemia, Pseudo-hypoglycemia and Severe and/or Confirmed Hypoglycemia) at Month 12
Description: Severe hypoglycemia: an event in which the child/adolescent having altered mental status and cannot assist in their care, is semiconscious or unconscious, or in coma ± convulsions and may require parenteral therapy (glucagon or glucose). Documented symptomatic hypoglycemia: an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of <=70 mg/dL (3.9 mmol/L). Asymptomatic hypoglycemia: an event not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose concentration <=70 mg/dL. Probable symptomatic hypoglycemia: an event during which symptoms of hypoglycemia were not accompanied by plasma glucose determination but was presumably caused by a plasma glucose concentration <=70 mg/dL. Pseudo-hypoglycemia:an event with any of the typical symptoms of hypoglycaemia with plasma glucose concentration >70 mg/dL.
Time Frame: Month 12
Population: Analysis was performed on the safety population which included all randomized participants who actually received who received at least 1 dose or part of a dose of IMP, and was analyzed according to treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 233 | 228
percentage of participants
  Any hypoglycemia | 99.1 | 98.7
  Severe Hypoglycemia | 8.6 | 11.0
  Documented Symptomatic Hypoglycemia | 94.8 | 93.9
  Probable Symptomatic Hypoglycemia | 10.3 | 13.6
  Asymptomatic Hypoglycemia | 88.4 | 89.5
  Pseudo-hypoglycemia | 15.9 | 14.5
  Severe and/or documented hypoglycemia | 99.1 | 98.2

11. Secondary Outcome: Percentage of Participants With Any Hyperglycemia With Ketosis at Month 12
Description: Hyperglycemia with ketosis was defined as SMPG >=252 mg/dL (14 mmol/L) with accompanying self-measured blood ketones >=1.5 mmol/L.
Time Frame: Month 12
Population: Analysis was performed on the safety population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 233 | 228
percentage of participants | 9.9 | 13.6

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form until the end of the study (Week 58) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are treatment-emergent adverse events that is AEs that developed, worsened or became serious during the 'on treatment period' (time from first dose of IMP up to 2 days after last injection of IMP). Analysis was performed on safety population.
Arm/Group | HOE901-U300 | Lantus
All-Cause Mortality (participants affected / at risk) | 1/233 | 0/228
Serious Adverse Events (participants affected / at risk) | 35/233 | 31/228
Other Adverse Events (participants affected / at risk) | 105/233 | 118/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HOE901-U300 (N=233) | Lantus (N=228)
Adrenal Insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Meningococcal Infection (Infections and infestations) | 0 (0) | 1 (1)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Electric Shock (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 3 (3) | 1 (1)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 5 (5) | 6 (6)
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Autonomic Nervous System Imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic Coma (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic Seizure (Nervous system disorders) | 8 (11) | 10 (10)
Hypoglycaemic Unconsciousness (Nervous system disorders) | 6 (10) | 10 (11)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anembryonic Gestation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Completed Suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1)
Testicular Torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HOE901-U300 (N=233) | Lantus (N=228)
Vomiting (Gastrointestinal disorders) | 14 (20) | 9 (10)
Gastroenteritis (Infections and infestations) | 12 (14) | 10 (14)
Influenza (Infections and infestations) | 14 (17) | 19 (25)
Nasopharyngitis (Infections and infestations) | 37 (57) | 39 (60)
Pharyngitis (Infections and infestations) | 14 (18) | 22 (29)
Upper Respiratory Tract Infection (Infections and infestations) | 20 (28) | 18 (21)
Ketosis (Metabolism and nutrition disorders) | 19 (50) | 30 (52)
Overweight (Metabolism and nutrition disorders) | 2 (2) | 13 (13)
Headache (Nervous system disorders) | 19 (38) | 15 (23)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 7 (7)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2016-08-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT02735044/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT02735044/SAP_001.pdf